CLINICAL TRIAL: NCT05688046
Title: Efficacy and Safety Analysis of Immune Checkpoint Inhibitors Plus Angiogenesis Inhibitors for Treatment of Advanced Driver-negative NSCLC in Elderly Patients：A Retrospective Study
Brief Title: Efficacy and Safety Analysis of ICIs Plus Angiogenesis Inhibitors for Treatment of Advanced NSCLC in Elderly Patients
Acronym: IMAGINE
Status: Completed | Type: Observational
Sponsor: Suzhou Municipal Hospital (Other)
Responsible Party: Principal Investigator, jing xue, Associate chief physician, Suzhou Municipal Hospital
Other Study IDs: IMAGINE
Record Dates: First submitted 2023-01-08; First posted 2023-01-18 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: NSCLC
Keywords: Elderly Patient
MeSH Terms: interventions — Immune Checkpoint Inhibitors; Angiogenesis Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- IA group: Immune checkpoint inhibitors plus angiogenesis inhibitors group
  Interventions: Drug: Immune checkpoint inhibitors plus angiogenesis inhibitors
- NIA group: Immune checkpoint inhibitors without angiogenesis inhibitors group
  Interventions: Drug: Immune checkpoint inhibitors without angiogenesis inhibitors

INTERVENTIONS:
Drug: Immune checkpoint inhibitors plus angiogenesis inhibitors — PD-(L)1-based therapy plus Bevacizumab or Anlotinib
  Groups: IA group
Drug: Immune checkpoint inhibitors without angiogenesis inhibitors — PD-(L)1-based therapy
  Groups: NIA group

SUMMARY:
Immune checkpoint inhibitors(ICIs) combined with angiogenesis inhibitors may is synergistic in elderly patients with advanced non-small cell lung cancer(NSCLC), however its true efficacy is still unclear. The investigators retrospectively compared clinical efficacy and safety of driver-negative elderly patients with advanced NSCLC treated with ICIs with(or without)angiogenesis inhibitors in the Cancer Center of the Affiliated Suzhou Hospital of Nanjing Medical University.

DETAILED DESCRIPTION:
The investigators reviewed the medical records of all lung cancer patients in the Cancer Diagnosis and Treatment Center of Suzhou Hospital Affiliated to Nanjing Medical University from January 1, 2019 to December 31, 2021, and a total of 79 patients were enrolled. The subjects were divided into two groups: the group treated with immune checkpoint inhibitors plus antiangiogenic drugs(IA group) and the group treated with immune checkpoint inhibitors without antiangiogenic drugs(NIA group). The data of PFS, OS, ORR, covariates, and Immune-related adverse events (irAEs) were collected through electronic medical records and follow-up. The primary endpoint of the study was PFS, and the secondary endpoints were OS, ORR and irAEs.All enrolled patients were followed up until August 1, 2022.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥65 years old.
2. Stage IV according to the AJCC Cancer grading manual (8th edition).
3. Histologically confirmed NSCLC.
4. No driver mutations.
5. Received at least 2 courses of immunotherapy.
6. Expected survival time > 3 months.
7. No concurrent malignancy.
8. Not participating in a clinical trial.
9. The functions of important organs were basically normal.
10. Sign informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The investigators retrospectively compared clinical efficacy and safety of driver-negative elderly patients with advanced NSCLC treated with ICIs with(or without)angiogenesis inhibitors in the Cancer Center of the Affiliated Suzhou Hospital of Nanjing Medical University.A total of 43 patients in the NIA group and 36 patients in the IA group were included in the study between January 1,2019 and December 31,2021.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
PFS | Up to August 1, 2022
  PFS was defined as the time from the start of the first immunotherapy until disease progression or death

SECONDARY OUTCOMES:
OS | Up to August 1, 2022
  OS was defined as the time from the start of the first immunotherapy to death from any cause
ORR | Up to August 1, 2022
  ORR refers to the sum of complete response and partial response to treatment
irAEs | Up to August 1, 2022
  Immune-related adverse events were evaluated according to the CTCAE5.0 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jing Xue, Principal Investigator — The Affiliated Suzhou Hospital of Nanjing Medical University
Locations (1):
- The Affiliated Suzhou Hospital of Nanjing Medical University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No